CLINICAL TRIAL: NCT03941431
Title: Optimally Sequential Treatment of Integrated Chinese and Western Medicine for Psoriasis: a Multicenter Randomized Controlled Trial
Brief Title: Sequential Treatment of Psoriasis With Integrated Traditional Chinese and Western Medicine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai Dermatology Hospital (Other); Chinese Medicine Hospital Affiliated to Southwest Medical University (Unknown); Wuhan No.1 Hospital (Other); The Second People's Hospital Affiliated to Fujian University of TCM (Unknown); Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1705304
Record Dates: First submitted 2019-05-01; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Jueyin granule; Moving cupping; NB-UVB; combination of Chinese traditional and Western medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chinese medicine internal treatment group (Experimental): Participants in Chinese medicine internal treatment group will receive Jueyin granule two times daily after meals and moving cupping placebo therapy three times per week for 8 weeks.
  Interventions: Drug: Jueyin granules; Device: moving cupping placebo therapy
- Chinese medicine external treatment group (Experimental): Participants in Chinese medicine internal treatment group will receive Jueyin placebo granule two times daily after meals and moving cupping therapy three times per week for 8 weeks.
  Interventions: Device: moving cupping therapy; Drug: Jueyin placebo granules
- Chinese medicine treatment group (Experimental): Participants in Chinese medicine treatment group will receive Jueyin granule two times daily after meals, moving cupping therapy and NB-UVB placebo therapy three times per week for 8 weeks.
  Interventions: Drug: Jueyin granules; Device: moving cupping therapy; Device: NB-UVB placebo phototherapy
- Western medicine treatment group (Experimental): Participants in Western medicine treatment group will receive Jueyin placebo granules two times daily after meals, moving cupping placebo therapy and NB-UVB therapy three times per week for 8 weeks.
  Interventions: Device: NB-UVB therapy; Drug: Jueyin placebo granules; Device: moving cupping placebo therapy
- Integrated Chinese and Western Medicine Treatment Group (Experimental): Participants in Chinese and Western Medicine Treatment Group will receive Jueyin granules two times daily after meals, moving cupping therapy and NB-UVB therapy three times per week for 8 weeks.
  Interventions: Drug: Jueyin granules; Device: moving cupping therapy; Device: NB-UVB therapy

INTERVENTIONS:
Drug: Jueyin granules — Jueyin granules p.o. once a day for 8 weeks.
  Other Names: Chinese Herbal Medicine
  Arms: Chinese medicine internal treatment group; Chinese medicine treatment group; Integrated Chinese and Western Medicine Treatment Group
Device: moving cupping therapy — Moving cupping therapy three times per week for 8 weeks.
  Arms: Chinese medicine external treatment group; Chinese medicine treatment group; Integrated Chinese and Western Medicine Treatment Group
Device: NB-UVB therapy — NB-UVB phototherapy three times per week for 8 weeks.
  Arms: Integrated Chinese and Western Medicine Treatment Group; Western medicine treatment group
Drug: Jueyin placebo granules — Jueyin placebo granules p.o. once a day for 8 weeks.
  Other Names: Chinese Herbal Medicine
  Arms: Chinese medicine external treatment group; Western medicine treatment group
Device: moving cupping placebo therapy — Moving cupping placebo therapy three times per week for 8 weeks.
  Arms: Chinese medicine internal treatment group; Western medicine treatment group
Device: NB-UVB placebo phototherapy — NB-UVB placebo phototherapy three times per week for 8 weeks.
  Arms: Chinese medicine treatment group

SUMMARY:
The purpose of this study was to explore intervention time of Chinese medicine and specification of a sequential treatment plan for severe psoriasis with Chinese and Western medicine.

DETAILED DESCRIPTION:
Psoriasis is a chronic, relapsing, inflammatory disease that seriously affects the quality of life of patients. Both Chinese medicine and Western medicine have many methods for treating psoriasis, each with its own advantages and disadvantages, but the pursuit of green and effective treatment programs is still the focus of the work of specialists and researchers. How to combine the existing safe and effective Chinese and Western medicine methods organically, and to achieve the purpose of improving efficacy under the premise of ensuring safety, is the motivation for carrying out this research.

The treatments involved in this study include cupping, phototherapy, and Chinese medicine. All three methods have sufficient literature to confirm their effectiveness in treating plaque psoriasis. The research team hopes to obtain a best combination of three treatments for plaque psoriasis by using a multicenter, randomized, single-blind, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Plaque psoriasis, the course of disease is not limited.
2. Skin lesions involving ≤ 15% BSA (the lesions are mainly located in the trunk and / or limbs, palm / sole, face / scalp, vulva area is not included).
3. 18 to 65 years old, male or female patient.
4. Informed consent must be obtained.

Exclusion Criteria:

1. other active skin diseases which may affect the condition assessment are present.
2. Patients who received systematic treatment of research drugs, biological agents and immunosuppressive agents within 2 months.
3. Patients who received treatment with topical glucocorticoids, phototherapy, etc. within 2 weeks.
4. Those with severe, uncontrollable local or systemic acute or chronic infections.
5. patients with severe systemic diseases; or clinical test indicators in one of the following cases: alanine transferase or glutamate transferase increased by >1.5 times the upper limit of normal; serum creatinine increased by >1.5 times the upper limit of normal Any of the main blood routine indicators (white blood cell count, red blood cell count, hemoglobin amount, platelet count) below the lower limit of normal; or other laboratory abnormalities judged by the investigator are not suitable for participation in this trial.
6. Patients with a history of malignant tumors and patients with primary or secondary immunodeficiency and hypersensitivity.
7. Patients underwent major surgery within 8 weeks or will require such surgery during the study period.
8. Patients who are pregnant or in lactation.
9. Those have a history of alcohol abuse, drug abuse or drug abuse.
10. Patients with a history of serious mental illness or family history.
11. Patients with a family history of cancer.
12. Other reasons that the investigator considered inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area and severity index | Up to 56 days after treatment.
  Psoriasis Area and Severity Index involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 56 days after treatment.
  The percentage of BSA involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%)
Physician Global Assessment (PGA) | Up to 56 days after treatment.
  Physician Global Assessment (PGA) is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), desquamation (D) across all psoriatic lesions. It is calculated as follows: PGA score = (E + I + D) / 3, then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0) - Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 56 days after treatment.
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 56 days after treatment.
  PRQoL is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 56 days after treatment.
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
TCM symptom score | Up to 56 days after treatment.
  The TCM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Department of dermatology, Shanghai Yueyang Integrated Medicine Hospital, Shanghai
Locations (6):
- China (6):
  - The Second People's Hospital Affiliated to Fujian University of TCM, Fuzhou, Fujian
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Chinese Medicine Hospital Affiliated to Southwest Medical University, Luzhou, Sichuan
  - Shanghai Dermatology Hospital, Shanghai
  - Shanghai Yueyang Integrated Medicine Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu Y, Sun X, Hu R, Xia P, Wei Y, Yang W, Huang N, Ding Y, Guo S, Yang C, Weng H, Zhang Y, Ding X, Huang Q, Zhou X, Li X, Li B. A Randomized Controlled Trial for the Optimal Implementation of Psoriasis Treatment by Integrating Chinese and Western Medicine. Psoriasis (Auckl). 2025 Mar 21;15:55-66. doi: 10.2147/PTT.S487536. eCollection 2025. PMID 40135074
- [Derived] Sun X, Zhou X, Wei Y, Yang W, Huang N, Ding Y, Hu R, Guo S, Yang C, Weng H, Zhang Y, Chen X, Ding X, Liu L, Yin Q, Wang R, Li X, Li B. Our Choice: study protocol for a randomized controlled trial for optimal implementation of psoriasis treatment by the integration of Chinese and western medicine. Trials. 2020 Mar 30;21(1):299. doi: 10.1186/s13063-020-4209-3. PMID 32228720